CLINICAL TRIAL: NCT04778618
Title: Impact of Optimal Doses of Antithymocyte Globulin Conditioning on Graft-versus- Host Disease and Virus Reactivation in Haploidentical Hematopoietic Stem Cell Transplantation
Brief Title: Individualized Dose Study of ATG in Haploidentical Hematopoietic Stem Cell Transplantation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Daihong Liu, Director, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2020-484-01
Record Dates: First submitted 2021-02-24; First posted 2021-03-03 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Haploidentical Hematopoietic Stem Cell Transplantation
MeSH Terms: interventions — Antilymphocyte Serum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Individual dose of Thymoglobulin (Experimental): Individual dose of Thymoglobulin (r-ATG) : Individual dose of ATG was Intravenous infused every day from day -5 to day -2 (total ATG dose was calculated based on pharmacokinetic index, within a range of 6 mg/kg to 10mg/kg)
  Interventions: Drug: Antithymocyte Globulin

INTERVENTIONS:
Drug: Antithymocyte Globulin — Individual dose of ATG was Intravenous infused every day from day -5 to day -2 (total ATG dose was calculated based on pharmacokinetic index, within a range of 6 mg/kg to 10mg/kg). Antithymocyte globulin (ATG) was added to conditioning regimens for 4 days (days -5 and -2). Prophylaxis against graft-versus-host disease (GVHD) was performed with cyclosporine A (CsA), mycophenolate mofetil (MMF) and short-term methotrexate

SUMMARY:
The purpose of this study is to determine the response and toxicity rate of two different dosages (Individualized dosage VS. fixed dosage) of ATG as a prophylaxis for acute GVHD in haploidentical peripheral blood stem cell transplantation (haplo-PBSCT).

DETAILED DESCRIPTION:
Acute graft-versus-host disease (aGvHD) is an important complication of haplo-HSCT. The Seattle group initially introduced the use of ATG as a treatment for acute graft-versus-host disease (aGVHD) in allogeneic hematopoietic stem cell transplantation (haplo-PBSCT) recipients. Presently, in both myeloablative and reduced-intensity conditioning (RIC) haplo-PBSCT, ATG is part of postengraftment immunosuppressive regimens.

The regimens for prophylaxis of GVHD based on 10mg/kg rabbit anti-human thymocyte immunoglobin (ATG, Thymoglobulin®, Genzyme Polyclonals S.A.S) effectively reduced the occurrence of grade II-IV aGvHD. However, the incidence of cytomegalovirus (CMV) and EB virus (EBV) reactivation were higher due to a slower immune reconstitution. The 100-day cumulative incidence of CMV and EBV viremia were both over 70% in our unmanipulated haplo-PBSCT program. The optimal dose of ATG balancing the efficacy of GVHD prophylaxis and the risk of virus reactivation in haplo-PBSCT remains unknown.

Reports on the pharmacokinetics of Thymoglobulin in allo-HSCT revealed a high variability. Recent pharmacokinetic studies have shown that the half-life of total ATG after transplant is longer than the active ATG (which is available to bind to human lymphocytes and causes the desired immunological effects). And active ATG appears more associated with pharmacodynamics effects. The investigators found that virus reactivation and acute GVHD were highly affected by ATG exposure (area under the curve, AUC) in previous cohort study. The investigators have found an optimal range of active ATG exposure balancing the efficacy of GVHD prophylaxis and the risk of virus reactivation. The incidence of CMV reactivation and III-IV aGVHD reduced to 60%, 6% respectively.

The results suggested that Individualized dosing of ATG has a potential advantage in balancing the efficacy of GVHD prophylaxis and the risk of virus reactivation in haplo-PBSCT. This may improve the survival and quality of life of patients undergoing haplo-PBSCT. A prospective randomized trial is required to compare the efficacy of Individualized dosage of ATG as a prophylaxis for acute GVHD in haplo-PBSCT.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of hematological malignancies refer to the 2016 WHO classification.
2. Aged 14 to 60 years.
3. Karnofsky or Lansky performance status [27] ≥ 70%. Please refer to Appendix A.
4. First transplantation.
5. Adequate organ function
6. Patient and/or legal guardian must sign informed consent for HSCT.

Exclusion Criteria:

1. Ex-vivo T-cell depleted grafts.
2. Pregnancy or breast-feeding or unwilling to use proper contraception.
3. Unable to assess whether the malignancy is in complete remission.
4. History of hypersensitivity to any biological product.
5. Sensibility to rabbit proteins or previous treatment with Thymoglobuline®.
6. Subjects with uncontrollable systemic infection (viral, bacterial or fungal).
7. Participation in other trial in which the dose of Thymoglobuline® is fixed other than individualized dose.
8. Unable to sign the informed consent form.

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 63 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2024-01-14 (Estimated)

PRIMARY OUTCOMES:
The cumulative incidences of CMV reactivation | 180 days after transplantation
  The cumulative incidences of CMV reactivation in participants after transplantation, tested by realtime PCR
The cumulative incidences of EBV reactivation | 180 days after transplantation
  The cumulative incidences of EBV reactivation in participants after transplantation, tested by realtime PCR

SECONDARY OUTCOMES:
Engraftment | 28 days after transplantation
  Neutrophil engraftment was defined as the first day with a neutrophil count > 0.5 × 10^9/L on three consecutive days postnadir; platelet engraftment was defined as the first day with a platelet count > 20 × 10^9/L without transfusion for five consecutive days postnadir.
The cumulative incidences of aGVHD (refer to MAGIC criteria) | 100 days after transplantation
  Defined as the proportion of participants who developed acute GVHD
The cumulative incidences of cGVHD (refer to NIH criteria) | 2 years after transplantation
  cGvHD was diagnosed and graded according to the 2014 National Institutes of Health (NIH) consensus criteria: mild, moderate or severe respectively.
Relapse | 1 years after transplantation
  Defined as reappearance of leukemic blasts in peripheral blood or ≥5% blasts in BM or reappearance or new appearance of extramedullary leukemia.
Nonrelapse mortality (NRM) | 1 years after transplantation
  Defined as death due to causes other than malignancy relapse
Disease-free survival (DFS) | 1 years after transplantation
  Defined as survival with no evidence of relapse or progression.
Overall survival (OS) | 1 year after transplantation
  Defined as the time from transplantation to last follow-up or death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Dai-hong Liu, Dr., Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Call SK, Kasow KA, Barfield R, Madden R, Leung W, Horwitz E, Woodard P, Panetta JC, Baker S, Handgretinger R, Rodman J, Hale GA. Total and active rabbit antithymocyte globulin (rATG;Thymoglobulin) pharmacokinetics in pediatric patients undergoing unrelated donor bone marrow transplantation. Biol Blood Marrow Transplant. 2009 Feb;15(2):274-8. doi: 10.1016/j.bbmt.2008.11.027. PMID 19167688
- [Background] Walker I, Panzarella T, Couban S, Couture F, Devins G, Elemary M, Gallagher G, Kerr H, Kuruvilla J, Lee SJ, Moore J, Nevill T, Popradi G, Roy J, Schultz KR, Szwajcer D, Toze C, Foley R; Canadian Blood and Marrow Transplant Group. Pretreatment with anti-thymocyte globulin versus no anti-thymocyte globulin in patients with haematological malignancies undergoing haemopoietic cell transplantation from unrelated donors: a randomised, controlled, open-label, phase 3, multicentre trial. Lancet Oncol. 2016 Feb;17(2):164-173. doi: 10.1016/S1470-2045(15)00462-3. Epub 2015 Dec 24. PMID 26723083
- [Background] Bacigalupo A, Lamparelli T, Barisione G, Bruzzi P, Guidi S, Alessandrino PE, di Bartolomeo P, Oneto R, Bruno B, Sacchi N, van Lint MT, Bosi A; Gruppo Italiano Trapianti Midollo Osseo (GITMO). Thymoglobulin prevents chronic graft-versus-host disease, chronic lung dysfunction, and late transplant-related mortality: long-term follow-up of a randomized trial in patients undergoing unrelated donor transplantation. Biol Blood Marrow Transplant. 2006 May;12(5):560-5. doi: 10.1016/j.bbmt.2005.12.034. PMID 16635791
- [Background] Bacigalupo A, Lamparelli T, Bruzzi P, Guidi S, Alessandrino PE, di Bartolomeo P, Oneto R, Bruno B, Barbanti M, Sacchi N, Van Lint MT, Bosi A. Antithymocyte globulin for graft-versus-host disease prophylaxis in transplants from unrelated donors: 2 randomized studies from Gruppo Italiano Trapianti Midollo Osseo (GITMO). Blood. 2001 Nov 15;98(10):2942-7. doi: 10.1182/blood.v98.10.2942. PMID 11698275
- [Background] Remberger M, Svahn BM, Mattsson J, Ringden O. Dose study of thymoglobulin during conditioning for unrelated donor allogeneic stem-cell transplantation. Transplantation. 2004 Jul 15;78(1):122-7. PMID 15257050
- [Derived] Wang H, Wang N, Wang L, Du J, Li F, Shao Y, Peng B, Luan S, Wang L, Jin X, Gao C, Dou L, Liu D. Targeted dosing of anti-thymocyte globulin in adult unmanipulated haploidentical peripheral blood stem cell transplantation: A single-arm, phase 2 trial. Am J Hematol. 2023 Nov;98(11):1732-1741. doi: 10.1002/ajh.27068. Epub 2023 Sep 14. PMID 37706580